CLINICAL TRIAL: NCT04598464
Title: Effect of Home-Based Exercise Program on Physical Function and Balance in Older Adults With Sarcopenia: A Multicenter Randomized Controlled Study
Brief Title: Effect of Home-Based Exercise Program in Older Adults With Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ekin Ilke Sen, Assistant Professor, Istanbul University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulU-2018-200
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The home-based training program
  Interventions: Other: Home based exercise
- control group (No Intervention): All patients participated in a one-session educational program conducted by the investigators at each clinic.

INTERVENTIONS:
Other: Home based exercise — The home-based training program included posture and stretching exercises, strengthening exercises, balance training, and a walking regimen 3 days per week for 3 months.
  Arms: Exercise group

SUMMARY:
In the prospective, randomized, controlled multi-centre study, 100 patients who were clinically diagnosed with sarcopenia were assigned to either a home-based exercise group or the control group. The home-based exercise program was performed three days per week for 12 weeks. Before and three months after the exercise program, all the patients were evaluated.

DETAILED DESCRIPTION:
Sarcopenia is a complex and multifactorial syndrome characterized by progressive and generalized loss of skeletal muscle mass and strength.The randomized, multicenter study was conducted at the physical medicine and rehabilitation departments of five different centers. One hundred patients met the inclusion and exclusion criteria and were randomly allocated to either a home-based exercise group (n=50) or a control group (n=50). The patients were evaluated before and 3 months after inclusion using the timed up and go test, the Berg balance scale, the 6-minute walk test , a numeric rating scale to determine QoL, and the number of falls.

ELIGIBILITY:
Inclusion Criteria:

community-dwelling older adult diagnosis of sarcopenia according to the clinical examination; and able to walk independently. The physical performance of patients with a SARC-F score ≥4 were tested using a gait speed test and a short physical performance battery (SPPB). The diagnosis of sarcopenia was confirmed in cases where the patient's gait speed was ≤0.8 m/s and the SPPB score was ≤8

Exclusion Criteria:

having cardiovascular, pulmonary, and/or chronic diseases that may affect participation in the exercise program; impaired cognition; previous diagnosis of a neurological condition that severely affected mobility and balance; malignancy; metastatic cancer; serious vision loss or vestibular impairment

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline timed up and go test at 3-months | Baseline, 3-month
  The timed up and go test test measures the amount of time needed for a patient to stand up from a chair, walk three meters as quickly and safely as possible toward a cone, walk around it, and sit down on the chair again.

SECONDARY OUTCOMES:
Change from baseline Berg balance scale score at 3-months | Baseline, 3-month
  The Berg balance scale is a reliable tool for assessing balance and postural control in older adults. This scale consists of 14 items, each scored from 0 to 4, with a maximal score of 56 points. A higher score indicates better balance
Change from baseline 6-minute walk test (6MWT) at 3-months | Baseline, 3-month
  The 6MWT is used to assess people's physical capacity. participants were asked to walk back and forth in a hospital corridor free of obstacles for 6 minutes at a regular pace.
Change from baseline self-reported QoL at 3-months | Baseline, 3-month
  The average level of QoL was evaluated using the numeric scale and scored between 0 and 10, where 0 indicates the best QoL and 10 indicates the worst QoL
Change from baseline number of falls at 3-months | Baseline, 3-month
  The number of falls was monitored by monthly telephone calls

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Karan, Professor, Principal Investigator — Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation
Locations (5):
- Turkey (Türkiye) (5):
  - Balikesir University Faculty of Medicine, Department of Physical Therapy and Rehabilitation, Balıkesir
  - Istanbul Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul
  - Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul
  - Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul
  - Ege University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sen EI, Eyigor S, Dikici Yagli M, Ozcete ZA, Aydin T, Kesiktas FN, Aydin FY, Vural M, Sahin N, Karan A. Effect of Home-Based Exercise Program on Physical Function and Balance in Older Adults With Sarcopenia: A Multicenter Randomized Controlled Study. J Aging Phys Act. 2021 Jul 16;29(6):1010-1017. doi: 10.1123/japa.2020-0348. PMID 34271551